CLINICAL TRIAL: NCT01899729
Title: A Randomized, Double-Blind, Placebo-Controlled, 12-week Dose-Ranging Trial of IMO-8400 in Patients With Moderate to Sever Plaque Psoriasis
Brief Title: A 12-week Dose-Ranging Trial in Patients With Moderate to Severe Plaque Psoriasis
Acronym: 8400-201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8400-201; 2013-000164-28 (EudraCT Number)
Record Dates: First submitted 2013-07-02; First posted 2013-07-15 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; autoimmune disease; Toll like receptor
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- IMO-8400 Regimen 1 (Experimental): IMO 8400 at 0.075 mg/kq q wk x 12 wks
  Interventions: Drug: IMO-8400 Regimen 1
- IMO-8400 Regimen 2 (Experimental): IMO-8400 at 0.15 mg/kg q wk x 12 wks
  Interventions: Drug: IMO-8400 Regimen 2
- IMO-8400 Regimen 3 (Experimental): IMO_8400 at 0.3 mg/kg q wk x 12 wks
  Interventions: Drug: IMO-8400 Regimen 3
- Placebo (Placebo Comparator): Saline (placebo) q wk x 12 wks
  Interventions: Drug: Saline Placebo
- IMO-8400 Regimen 4 (Experimental): IMO_8400 at 0.6 mg/kg q wk x 12 wks
  Interventions: Drug: IMO-8400 Regimen 4

INTERVENTIONS:
Drug: IMO-8400 Regimen 1 — IMO-8400 0.075 mg/kg q wk x 12 wk by subcutaneous injection
  Arms: IMO-8400 Regimen 1
Drug: IMO-8400 Regimen 2 — IMO-8400 0.15 mg/kg q wk x 12 wk by subcutaneous injection
  Arms: IMO-8400 Regimen 2
Drug: IMO-8400 Regimen 3 — IMO-8400 0.3 mg/kg q wk x 12 wk by subcutaneous injection
  Arms: IMO-8400 Regimen 3
Drug: Saline Placebo — Saline q wk x 12 wk by subcutaneous injection
  Arms: Placebo
Drug: IMO-8400 Regimen 4 — IMO-8400 0.6 mg/kg q wk x 12 wk by subcutaneous injection
  Arms: IMO-8400 Regimen 4

SUMMARY:
IMO 8400 is a second-generation oligonucleotide antagonist of endosomal Toll-like receptors (TLR) 7, TLR8 and TLR9. These TLR react to complexes of exogenous nucleic acids (as might be encountered during infection) and endogenous nucleic acids (as might be released during tissue damage during autoimmune disease). In vitro and in multiple animal models of autoimmune disease, IMO-8400 blocks immune activation mediated through TLR7, 8 and 9. In Phase 1 studies (Protocol 8400-001) IMO 8400 has been administered to healthy adults by SC injection at single-doses and multiple-doses (4 weeks) up to 0.6 mg/kg. All treatments were well-tolerated, with mild injection site reactions and no pattern of systemic reactions or laboratory changes.

The current study represents the first clinical trial of IMO-8400 in patients with active autoimmune disease. Moderate to severe plaque psoriasis was chosen for this 12-week proof of activity trial based on a prior 4-week study using a first generation TLR7 and 9 antagonist which demonstrated clinical improvement in this patient population.

DETAILED DESCRIPTION:
Eligible subjects will be enrolled and randomized to receive one of the four treatments (three dose levels of IMO-8400 or Saline Placebo). Treatments will be administered once weekly by subcutaneous injections. Subjects will received treatment for 12 weeks and then be followed for an additional 6 weeks to assess the durability of the response.

ELIGIBILITY:
Inclusion Criteria:

1. Is age 18 to 70 years, inclusive
2. Completes the informed consent procedure (see Section 15.2), including signing and dating the informed consent form
3. Has moderate to severe plaque psoriasis meeting the criteria specified above
4. Is willing and able to comply with the restrictions detailed above
5. Female subjects must have a negative pregnancy test at screening and on Day 1 prior to start of treatment
6. Female subjects of childbearing potential (see Section 8.2) and male subjects who have partners of childbearing potential must agree to use effective birth control (contraception; see Section 8.2) from Screening through the treatment period and for ninety (90) days after the last injection of study drug

Exclusion Criteria:

1. Has known hypersensitivity to any oligodeoxynucleotide
2. Is nursing
3. Has body weight <50 kg
4. Has BMI >34.9 kg/m2
5. Regularly consumes >3 drinks of alcoholic beverages (beer, wine, or distilled spirits) per day
6. Has a positive test for antibody to human immunodeficiency virus (HIV-1 or -2) or hepatitis C virus (HCV)
7. Has a positive test for hepatitis B surface antigen (HBsAg)
8. Has at screening safety laboratory tests meeting one or more of the following criteria:

   * hemoglobin <6.52 mmol/L (<10.5 g/dL)
   * white blood cell count <4x109/L ( <4,000/mm3)
   * absolute neutrophil count (ANC) <1.5x109/L (<1500/mm3)
   * platelet count <100x109/L (<100,000/mm3 )
   * serum creatinine >1.3x ULN;
   * alanine transaminase (ALT; SGPT) >2.5x ULN
   * aspartate transaminase (AST; SGOT) >2.5x ULN
   * serum total bilirubin >1.4x ULN (except if consistent with Gilbert's disease: i.e., total bilirubin <103 μmol/L (6 mg/dL) and conjugated bilirubin <1.2x ULN)
9. Has a history of allogeneic organ transplant (including bone marrow or stem cells)
10. Has, within the past 10 years, had evidence of or required treatment for cancer (except for treated, non-invasive carcinoma of the skin or cured cervical carcinoma-in-situ)
11. Has had within the past three months or is expected to have during the study period any of the following treatments:

    * surgery requiring general anesthesia
    * hematopoietic stimulating agents (e.g., erythropoietin, G-CSF, GM-CSF)
    * another investigational drug;
12. Has other significant medical conditions (chronic or active within the past 6 months), including, but not limited to: cardiac disease (e.g., unstable angina, myocardial infarction, congestive heart failure, ventricular arrhythmia); uncontrolled seizure disorder; liver disease; uncontrolled diabetes
13. Has any other condition that would, in the opinion of the Investigator, potentially compromise the safety or compliance of the patient or may preclude the patient's successful completion of the clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koos J Burggraaf, MSc, MD, PhD, Principal Investigator — Center Human Drug Research, Leiden, Netherlands
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

REFERENCES:
- [Derived] Balak DM, van Doorn MB, Arbeit RD, Rijneveld R, Klaassen E, Sullivan T, Brevard J, Thio HB, Prens EP, Burggraaf J, Rissmann R. IMO-8400, a toll-like receptor 7, 8, and 9 antagonist, demonstrates clinical activity in a phase 2a, randomized, placebo-controlled trial in patients with moderate-to-severe plaque psoriasis. Clin Immunol. 2017 Jan;174:63-72. doi: 10.1016/j.clim.2016.09.015. Epub 2016 Nov 20. PMID 27876460

RESULTS

PARTICIPANT FLOW:
Groups:
- IMO-8400 Regimen 1: IMO-8400 at 0.075 mg/kq q wk x 12 wks
  IMO-8400 Regimen 1: IMO-8400 0.075 mg/kg q wk x 12 wk by subcutaneous injection
- IMO-8400 Regimen 3: IMO-8400 at 0.3 mg/kg q wk x 12 wks
  IMO-8400 Regimen 3: IMO-8400 0.3 mg/kg q wk x 12 wk by subcutaneous injection
- IMO-8400 Regimen 4: IMO-8400 at 0.6 mg/kg q wk x 12 wk by subcutaneous injection
Period: Overall Study
Arm/Group | IMO-8400 Regimen 1 | IMO-8400 Regimen 2 | IMO-8400 Regimen 3 | IMO-8400 Regimen 4 | Placebo
Started | 9 | 9 | 8 | 9 | 11
Completed | 7 | 7 | 6 | 9 | 9
Not Completed | 2 | 2 | 2 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | IMO-8400 Regimen 1 | IMO-8400 Regimen 2 | IMO-8400 Regimen 3 | IMO-8400 Regimen 4 | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 11 | 46
Age, Continuous [Median (Full Range); unit: years] | 53 [19 to 66] | 31 [20 to 66] | 42.5 [20 to 70] | 45 [23 to 65] | 44 [25 to 66] | 44 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 1 | 2 | 12
  Male | 5 | 6 | 6 | 8 | 9 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 8 | 6 | 9 | 8 | 36
  More than one race | 2 | 0 | 0 | 0 | 1 | 3
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Netherlands | 9 | 9 | 8 | 9 | 11 | 46
Body Mass Index [Median (Full Range); unit: kg/m^2] | 26.5 [18.0 to 31.8] | 21.2 [19.2 to 33.8] | 27.15 [25.2 to 28.6] | 27.7 [19.6 to 40.4] | 30.9 [25.3 to 36.1] | 27.2 [18.0 to 40.4]

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of IMO-8400 Compared With Placebo
Description: The number of adverse events related and not related to treatment
Time Frame: 19 weeks (12 weeks on treatment + 7 week follow up)
Population: Safety population
Measure: Number; unit: adverse events
Groups:
- IMO-8400 Regimen 2: IMO-8400 at 0.15 mg/kg q wk x 12 wks IMO-8400 Regimen 2: IMO-8400 0.15 mg/kg q wk x 12 wk by subcutaneous injection
- Placebo: Saline (placebo) q wk x 12 wks
  Saline Placebo:
  Saline q wk x 12 wk by subcutaneous injection
Arm/Group | IMO-8400 Regimen 1 | IMO-8400 Regimen 2 | IMO-8400 Regimen 3 | IMO-8400 Regimen 4 | Placebo
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 11
adverse events
  AE Related to Treatment | 6 | 6 | 6 | 5 | 6
  AE Not Related to Treatment | 3 | 3 | 2 | 4 | 5
Statistical Analysis 1: Comparison: IMO-8400 Regimen 1 vs IMO-8400 Regimen 2 vs IMO-8400 Regimen 3 vs IMO-8400 Regimen 4 vs Placebo; Test type: Other — Used mixed effects model; p = 0.06, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to Study Day 113.
Description: An Adverse Event is any untoward medical occurrence temporally associated with the use of a medical product in a subject, whether or not the event is considered causally related to the medical product. An AE can be a new occurrence or an existing process that increases significantly in intensity or frequency.
Arm/Group | IMO-8400 Regimen 1 | IMO-8400 Regimen 2 | IMO-8400 Regimen 3 | IMO-8400 Regimen 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/8 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/8 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 8/9 | 8/9 | 7/8 | 7/9 | 9/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMO-8400 Regimen 1 (N=9) | IMO-8400 Regimen 2 (N=9) | IMO-8400 Regimen 3 (N=8) | IMO-8400 Regimen 4 (N=9) | Placebo (N=11)
Influenza like illness (General disorders) | 1 | 3 | 2 | 1 | 1
Injection site hematoma (General disorders) | 1 | 2 | 3 | 1 | 2
Fatigue (General disorders) | 1 | 3 | 1 | 1 | 1
Injection site pruritis (General disorders) | 1 | 1 | 1 | 0 | 0
Injection site pain (General disorders) | 2 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 2 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 2 | 4 | 5
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes